CLINICAL TRIAL: NCT06433427
Title: Metabolic Dysregulation as Biomarker of Frailty: Role of the Mitochondrial Dysfunction
Acronym: FRAMITO
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital of Ferrara (Other)
Collaborators: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Other Study IDs: 653/2023/Oss/AOUFe
Record Dates: First submitted 2024-03-14; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-01

CONDITIONS: Aging; Frailty; Mitochondrial Dysfunction; Chronic Disease
Keywords: Metabolic dysregulation
MeSH Terms: conditions — Frailty; Mitochondrial Diseases; Chronic Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — The laboratory of Oncology and Molecular Pathology of the University of Milano Bicocca will perform DNA extraction and the mtDNA damage evaluation by Real Time PCR analysis on PBMCs and sorted T and B lymphocytes and monocytes, obtained from each participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Non-Frail without Multimorbidity (NFWoM): Individuals aged 65 years or older without frailty and without multimorbidity. This group will serve as a reference for participants who are not frail and do not have multiple chronic conditions.
- Frail with Multimorbidity (FWM): Frail individuals aged 65 years or older who have multimorbidity. This group will include participants who exhibit frailty and have two or more chronic diseases.
- Frail without Multimorbidity (FWoM): Frail individuals aged 65 years or older without multimorbidity. This group will help assess frailty in the absence of multiple chronic conditions.

SUMMARY:
The goal of this observational study is to evaluate the presence of mitochondrial dysfunction related to oxidative stress and its possible role in frailty, with and without multimorbidity, and to identify possible frailty biomarkers correlated with mitochondrial dysfunction. The main questions it aims to answer are:

* What is the role of oxidative stress-related mitochondrial dysfunction in frailty, taking into account the interaction with multimorbidity.
* What could be the specific biomarkers associated with mitochondrial dysfunction in the assessment of frailty.

In order to reach the study goals, we will enroll three categories of older adults:

* Non-Frail without Multimorbidity (NFWoM);
* Frail with Multimorbidity (FWM);
* Frail without Multimorbidity (FWoM).

Each individual will undergo an assessment of frailty phenotype and multimorbidity, and the collection of blood samples to isolate Peripheral Blood Mononuclear Cells (PBMCs). The identification of frailty biomarkers in each group of participants will be performed by combining untargeted metabolomics-based approaches and functional studies on specific mitochondrial dysfunctions performed on PBMCs and their subpopulations. Multivariate statistical and machine learning techniques will characterize the three clinical phenotype groups based on molecular data.

DETAILED DESCRIPTION:
Study type: observational prospective study. Primary aim: is to evaluate the presence of mitochondrial dysfunction related to oxidative stress and its possible role in frailty, with and without multimorbidity.

Primary endpoint: mitochondrial dysfunction in frailty. Secondary aims: to combine untargeted metabolomics-based approaches and functional studies on specific mitochondrial dysfunctions performed on PBMCs and PBMC subpopulations (B lymphocytes, T lymphocytes and monocytes).

The research activities are organized in the following tasks:

* Task 1, Patient Enrollment: We will enroll individuals aged 65 years or older from geriatric outpatient clinics or geriatric wards. For each individual, we will perform an assessment of frailty and multimorbidity, and collect blood samples to isolate Peripheral Blood Mononuclear Cells (PBMCs). Three categories of individuals will be enrolled: 25 non-frail individuals without multimorbidity (NFWoM), 25 frail individuals with multimorbidity (FWM), and 25 frail individuals without multimorbidity (FWoM).
* Task 2, Separation of PBMC Subpopulations: T lymphocytes, B lymphocytes, and monocytes will be separated from frozen PBMCs using the Cell Sorting Facility for Fluorescence-Activated Cell Sorting (FACS) separation and the MoFlo Astrios cell sorter. The analyses on CD45+/CD3+/CD19-/CD14- T lymphocytes, CD45+/CD3-/CD19+/CD14- B lymphocytes, CD45+/CD3-/CD19-/CD14+ monocytes.
* Task 3, Mitochondrial Dysfunction Analysis on PBMCs and PBMC Subpopulations: For each individual, mitochondrial dysfunction will be evaluated by analyzing mtDNA damage (by Real-Time PCR), mitochondrial mass alteration (by Mitotracker staining), and intracellular and mitochondrial Reactive Oxygen Species (by DCF and MitoSOX staining). Moreover, we will evaluate alteration of glycolytic and mitochondrial metabolism using Agilent Seahorse Extracellular Flux Analyzer XFe96.
* Task 4, Untargeted Metabolomics on PBMCs and PBMC Subpopulations: To assess metabolic signature of PBMCs and subpopulations and highlight metabolic dysregulations linked to frailty, we will perform untargeted LC-MS-based metabolomics on PBMCs, T lymphocytes, B lymphocytes, and monocytes. The analysis on the polar metabolome will allow us to understand better the metabolic alterations associated with mitochondrial dysregulation.
* Task 5, Characterization of Biomarkers and Molecular Mechanism of Frailty: The potential biomarkers of frailty and the molecular mechanisms involved in mitochondrial dysfunction will be studied using statistical and machine learning techniques on molecular, metabolic and clinical data. This step will help characterize clinical phenotypes based on molecular measurements.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years
* Stable clinical conditions
* Willingness to participate in the study (provision of informed consent)
* Proficiency in the Italian language

Exclusion Criteria:

- Acute or unstable clinical conditions

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: The study will enroll individuals aged 65 years or older. The enrollment will take place among patients accessing geriatric outpatient clinics or being discharged from geriatric wards in clinically stable conditions.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2024-05-29 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2026-02-22 (Estimated)

PRIMARY OUTCOMES:
Difference in the mtDNA copy number between frail individuals with vs without multimorbidity | Baseline
  mtDNA copies isolated from total PBMCs and from T and B lymphocytes and monocytes, obtained from the participants, with JetQuick™ Blood and Cell Culture DNA Midiprep Kit (Invitrogen), and 10 ng of DNA will be used for analysis on QuantumStudio 7 Real Time PCR (Applied Biosystems). mtDNA copy number will be calculated by normalising the mitochondrial ND1 gene (mtND1) levels to nuclear Beta-2 microglobulin (B2M) levels.
  The number mtDNA copies will be compared between individuals with frailty and multimorbidity vs individuals with frailty without multimorbidity. Frailty will be derived based on the presence of at least three criteria among: involuntary weight loss ≥ 4.5 kg, muscle weakness measured by handgrip, self-reported fatigue on ≥ 3 days per week, low physical activity (assessed with the IPAQ questionnaire), and reduced gait speed (measured by the 4-m walking test). Multimorbidity will be defined as the presence of at least two chronic diseases.
Difference in the mtDNA copy number between non-frail vs frail individuals without multimorbidity | Baseline
  mtDNA copies isolated from total PBMCs and from T and B lymphocytes and monocytes, obtained from the participants, with JetQuick™ Blood and Cell Culture DNA Midiprep Kit (Invitrogen), and 10 ng of DNA will be used for analysis on QuantumStudio 7 Real Time PCR (Applied Biosystems). mtDNA copy number will be calculated by normalising the mitochondrial ND1 gene (mtND1) levels to nuclear Beta-2 microglobulin (B2M) levels.
  The number mtDNA copies will be compared between individuals with frailty and multimorbidity vs individuals with frailty without multimorbidity. Frailty will be derived based on the presence of at least three criteria among: involuntary weight loss ≥ 4.5 kg, muscle weakness measured by handgrip, self-reported fatigue on ≥ 3 days per week, low physical activity (assessed with the IPAQ questionnaire), and reduced gait speed (measured by the 4-m walking test). Multimorbidity will be defined as the presence of at least two chronic diseases.

SECONDARY OUTCOMES:
Variation in the mean intensity of mitochondrial fluorescence between non-frail vs frail individuals without multimorbidity | Baseline
  500,000 PBMCs obtained from the study participants will be stained with CD45, CD3, CD19 and CD14 antibodies and incubated with 100 nM Mitotracker Deep Red (Thermo Fisher Scientific) for 30 minutes at 30°C. Cells will be also labelled with Live/Dead dye and analyzed by flow cytometry with MoFLO Astrios cell sorter. Mitochondrial mass, evaluated as the median fluorescence intensity (MFI) of Mitotracker Deep Red, will be assessed in total PBMCs, T and B lymphocytes and monocytes. 40,000 events in each population gate will be acquired and offline analysis will be performed with Kaluza software.
Variation in the mean intensity of mitochondrial fluorescence between frail individuals with vs without multimorbidity | Baseline
  500,000 PBMCs obtained from the study participants will be stained with CD45, CD3, CD19 and CD14 antibodies and incubated with 100 nM Mitotracker Deep Red (Thermo Fisher Scientific) for 30 minutes at 30°C. Cells will be also labelled with Live/Dead dye and analyzed by flow cytometry with MoFLO Astrios cell sorter. Mitochondrial mass, evaluated as the median fluorescence intensity (MFI) of Mitotracker Deep Red, will be assessed in total PBMCs, T and B lymphocytes and monocytes. 40,000 events in each population gate will be acquired and offline analysis will be performed with Kaluza software.
Difference of intracellular Reactive Oxygen Species (ROS) between non-frail vs frail individuals without multimorbidity | Baseline
  The fluorescent cell-permeable indicator 2',7'-dichlorofluorescin diacetate (DCFH-DA) will be used for detecting intracellular ROS. DCFH-DA is deacetylated by cellular esterases to a non-fluorescent compound, which is later oxidised by ROS into fluorescent 2',7'-dichlorofluorescein (DCF). The intensity of the generated fluorescent signal correlates with the intracellular level of ROS. 500,000 PBMCs obtained from 25 NFWoM, 25 FWM and 25 FWoM subjects will be stained with CD45, CD3, CD19 and CD14 antibodies and incubated with 10 μM 2',7'-dichlorofluorescin diacetate (DCFH-DA) at 37°C for 30 minutes. Cells will be also labelled with Live/Dead dye and analyzed by flow cytometry. Intracellular ROS, evaluated as the median fluorescence intensity (MFI) of DCF, will be assessed in total PBMCs, T and B lymphocytes and monocytes. 40,000 events in each population gate will be acquired and offline analysis will be performed with Kaluza software.
Difference of intracellular Reactive Oxygen Species (ROS) between frail individuals with vs without multimorbidity | Baseline
  The fluorescent cell-permeable indicator 2',7'-dichlorofluorescin diacetate (DCFH-DA) will be used for detecting intracellular ROS. DCFH-DA is deacetylated by cellular esterases to a non-fluorescent compound, which is later oxidised by ROS into fluorescent 2',7'-dichlorofluorescein (DCF). The intensity of the generated fluorescent signal correlates with the intracellular level of ROS. 500,000 PBMCs obtained from 25 NFWoM, 25 FWM and 25 FWoM subjects will be stained with CD45, CD3, CD19 and CD14 antibodies and incubated with 10 μM 2',7'-dichlorofluorescin diacetate (DCFH-DA) at 37°C for 30 minutes. Cells will be also labelled with Live/Dead dye and analyzed by flow cytometry. Intracellular ROS, evaluated as the median fluorescence intensity (MFI) of DCF, will be assessed in total PBMCs, T and B lymphocytes and monocytes. 40,000 events in each population gate will be acquired and offline analysis will be performed with Kaluza software.
Qualitative difference in metabolomics profiles of PBMCs and PBMC subpopulations between non-frail vs frail individuals without multimorbidity | Baseline
  Untargeted LC-MS-based metabolomics will be performed on PBMCs and on T and B lymphocytes and monocytes, obtained as described in Task 2. Cell samples will be quenched using cold methanol. After protein precipitation, metabolites will be extracted and analysed by liquid chromatography mass spectrometry (LC-MS). Hydrophilic interaction chromatography (HILIC) will be used to resolve the polar metabolome before MS detection using an Agilent 6546 lc/q-tof instrument (Agilent).The whole protein content will be quantified with NanoDrop™ (Thermofisher) and used to normalize the metabolic profile of each sample.
Qualitative difference in metabolomics profiles of PBMCs and PBMC subpopulations between frail individuals with vs without multimorbidity | Baseline
  Untargeted LC-MS-based metabolomics will be performed on PBMCs and on T and B lymphocytes and monocytes, obtained as described in Task 2. Cell samples will be quenched using cold methanol. After protein precipitation, metabolites will be extracted and analysed by liquid chromatography mass spectrometry (LC-MS). Hydrophilic interaction chromatography (HILIC) will be used to resolve the polar metabolome before MS detection using an Agilent 6546 lc/q-tof instrument (Agilent).The whole protein content will be quantified with NanoDrop™ (Thermofisher) and used to normalize the metabolic profile of each sample.

CONTACTS AND LOCATIONS:
Overall Officials: Caterina Trevisan, PhD, Principal Investigator — Università degli Studi di Ferrara

REFERENCES:
- [Derived] Locatelli E, Torsello B, De Marco S, Lombardi M, Remelli F, Pampolini G, Ferrighi E, Bursi M, Bellotti A, Pasquale V, Ducci G, Navaei O, Candeloro R, Ferrara MC, Guo W, Cucini E, Bellelli G, Castellazzi M, Sacco E, Paglia G, Mazzola P, Bernasconi DP, Bianchi C, Trevisan C. Mitochondrial dysfunction as a biomarker of frailty: The FRAMITO study protocol. Arch Gerontol Geriatr. 2025 Jun;133:105803. doi: 10.1016/j.archger.2025.105803. Epub 2025 Feb 26. PMID 40043348